CLINICAL TRIAL: NCT06114641
Title: Effectiveness & Safety of Ovine Enoxaparin Sodium to Originator Enoxaparin in Non-ST-Segment Elevation ACS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENOX-0422
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Safety Issues; Effect of Drug
MeSH Terms: interventions — enoxaparin sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): Initial dose 30 mg IV loading dose is administered and followed by 1 mg/kg subcutaneously every 12 hours
  Interventions: Drug: Enoxaparin sodium injection
- Comparator (Active Comparator): Initial dose 30 mg IV loading dose is administered and followed by 1 mg/kg subcutaneously every 12 hours
  Interventions: Drug: Enoxaparin sodium injection

INTERVENTIONS:
Drug: Enoxaparin sodium injection — Originator Enoxaparin with a trade name is Lovenox.
  Other Names: Originator Enoxaparin

SUMMARY:
The aim of this study is evaluating safety and effectiveness of Ovine Enoxaparin Sodium in Non-ST-Segment Elevation Acute Coronary Syndrome (NSTEACS) Patients

DETAILED DESCRIPTION:
To assess the non-inferiority of Ovine Enoxaparin Sodium compared to Originator enoxaparin on the proportion of death, recurrent or refractory angina, and stroke during hospitalization within 10 days.

Effectiveness:

● Number and percentage of subjects with the composite of major adverse cardiac events (MACE) including death, recurrent myocardial infarction, recurrent angina, stroke, and unplanned revascularization after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30 days post initial administration.

Safety:

* Number and percentage of subjects with major bleeding occurring after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days using BARC scoring system.
* Number and percentage of subjects with minor bleeding occurring after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days using BARC scoring system.
* Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-3 post initial administration.
* Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-6 post initial administration.
* Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-10(+7) post initial administration.
* Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration at 30(+10) days post initial administration
* Number and percentage of subjects with any serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days.
* Number and percentage of subjects with any serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30(+10) days post initial administration.
* Number and percentage of subjects with non-serious adverse events after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30(+10) days post initial administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of non-ST-segment Elevation Acute Coronary Syndrome (NSTEACS) (unstable angina pectoris or Non-ST-Segment-Elevation myocardial infarction (NSTEMI)) based on particular diagnosis criteria
* Subjects with a diagnosis of non-ST-segment Elevation Acute Coronary Syndrome (NSTEACS) (unstable angina pectoris or Non-ST-Segment-Elevation myocardial infarction (NSTEMI)) based on particular diagnosis criteria
* Subjects or legally acceptable representatives have been informed properly regarding the study and signed the informed consent form

Exclusion Criteria:

* Subject concomitantly enrolled or scheduled to be enrolled in another study.
* Subjects use any other anticoagulant agent.
* Hemoglobin level below or equal to 9 mg/dl (for male) and 8.5 mg/dl (for female) or active bleeding.
* Any severe hematologic disease or history of intracerebral mass, aneurysm, arteriovenous malformation, recent (<6 months) ischemic stroke or TIA, recent (< 6 months) intracranial hemorrhage or gastrointestinal or genitourinary bleeding within the past 2 weeks.
* History of allergy or hypersensitivity to enoxaparin heparin or its derivatives, including other low molecular weight heparins (LWMH).
* History of Heparin type II-induced thrombocytopenia (HIT).
* Have severe renal failure (Creatinine Clearance below 15 mL/min), acute infectious endocarditis, hemodynamic instability, life threatening arrhythmia and cardiac arrest.
* A recent (<48 hours) or under spinal/epidural anesthesia.
* Platelet count below or equal to 100,000/mm3 at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
The non-inferiority of Ovine Enoxaparin Sodium compared to Originator enoxaparin on the proportion of death, recurrent or refractory angina, and stroke during hospitalization | During hospitalization or maximum within 10 days.
  Number and precentage non-inferiority of Ovine Enoxaparin Sodium compared to Originator enoxaparin on the proportion of death, recurrent or refractory angina, and stroke during hospitalization

SECONDARY OUTCOMES:
The composite of MACE including death, recurrent myocardial infarction, recurrent angina, stroke, and unplanned revascularization after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30 days post initial administration. | Within 30 days post initial administration.
  Number and precentage of the subjects with the composite of major adverse cardiac events (MACE) including death, recurrent myocardial infarction, recurrent angina, stroke, and unplanned revascularization after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30 days post initial administration.
The major bleeding after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days using BARC scoring system during hospitalization or maximum within 10 days. | During hospitalization or maximum within 10 days.
  Number and precentage of subjects with major bleeding after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days.
The minor bleeding after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days. | During hospitalization or maximum within 10 days.
  Number and precentage of subjects with the minor bleeding after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days.
The thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-3 post initial administration | Day-3 post initial administration
  Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-3 post initial administration
The thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-6 post initial administration | Day-6 post initial administration
  Number and precentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-6 post initial administration
The thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-10(+7) post initial administration | Day-10(+7) post initial administration
  Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on day-10(+7) post initial administration
The thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on 30(+10) days post initial administration | 30(+10) days post initial administration
  Number and percentage of subjects with thrombocytopenia events after Ovine Enoxaparin Sodium and Originator enoxaparin administration on 30(+10) days post initial administration
Serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration during hospitalization or maximum within 10 days During hospitalization or maximum within 10 days. | During hospitalization or maximum within 10 days.
  Number and percentage of subjects with any serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration During hospitalization or maximum within 10 days
Serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration on 30(+10) days post initial administration. | 30(+10) days post initial administration.
  Number and percentage of subjects with any serious adverse event after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30(+10) days post initial administration on 30(+10) days post initial administration.
Non-serious adverse events after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30(+10) days post initial administration. | 30(+10) days post initial administration.
  Number and percentage of subjects with non-serious adverse events after Ovine Enoxaparin Sodium and Originator enoxaparin administration within 30(+10) days post initial administration.

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Widyantoro, Ph.D, Principal Investigator — Indonesian Heart Association
Locations (3):
- Indonesia (3):
  - RSUP Dr.Sardjito, Yogyakarta, Yogyakarta, D.I.Yogyakarta
  - RS Jantung dan Pembuluh Darah Harapan Kita, Jakarta, Jakarta, DKI Jakarta
  - RSUP Prof. Dr. I.G.N.G Ngoerah, Bali, Bali